CLINICAL TRIAL: NCT02151877
Title: Efficacy of Nitric Oxide Administration in Attenuating Ischemia/Reperfusion Injury During Neonatal Cardiopulmonary Bypass.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Mallinckrodt (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: K5900209
Record Dates: First submitted 2014-05-27; First posted 2014-06-02 (Estimated); Results first posted 2020-04-03 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Ischemia/Reperfusion Injury After Neonatal Cardiac Surgery; Inflammatory Reaction After Neonatal Cardiac Surgery
Keywords: Ischemia/reperfusion injury
MeSH Terms: conditions — Ischemia; Reperfusion Injury | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nitric oxide on CPB (Experimental): neonates receiving inhaled NO into the cardiopulmonary bypass circuit during cardiac surgery
  Interventions: Drug: Inhaled Nitric Oxide
- control (Placebo Comparator): neonates not receiving inhaled NO into the cardiopulmonary bypass
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Inhaled Nitric Oxide — delivering inhaled Nitric Oxide into the cardiopulmonary bypass circuit during neonatal cardiac surgery
  Other Names: study group
  Arms: Nitric oxide on CPB
Drug: placebo — inhaled Nitric Oxide not delivered to the cardiopulmonary bypass circuit during neonatal cardiac surgery
  Other Names: control group
  Arms: control

SUMMARY:
Around 7500 neonates born yearly in the United States have complex congenital heart disease that require surgical repair in the first few days of life. The complexity of the surgical repair requires long periods of cardiopulmonary bypass (CPB) and the use of intermittent periods of low flow or complete circulatory arrest. The immature neonatal vital organs are more prone to the complications of the cardiopulmonary bypass circulation, namely ischemia/reperfusion (I/R) injury and systemic inflammatory response. Inhaled nitric oxide (NO) is used frequently in neonates for the treatment of pulmonary hypertension, Additionally, many studies have shown that NO has an anti-inflammatory effect by reducing I/R injury and endothelial dysfunction.

The purpose of this pilot study is to assess the efficacy of NO administration via the CPB circuit in attenuating the CPB induced I/R injury and systemic inflammatory reaction in neonates undergoing repair of complex congenital heart defects. Specific goals will be to demonstrate that NO use via CPB will:

* Decrease markers of I/R injury and systemic inflammatory response.
* Decrease platelet activation leading to reduced postoperative bleeding and transfusion requirements.
* Decrease postoperative organ dysfunction, and hence decrease operative mortality and postoperative morbidity.

Twelve neonates undergoing repair of complex congenital heart defects will receive NO via the CPB circuit, for the duration of surgery. They will be compared to a control group of 12 similar patients. Serum levels of different ischemic reperfusion injury and inflammatory markers will be measured at different time points after surgery and will be correlated with different end organ function tests and clinical course in the postoperative period. The results will be compared between the two groups to try to determine the clinical benefit of NO administration through CPB circuit.

ELIGIBILITY:
Inclusion Criteria:

* Neonates, age 0-30 days
* Full term, > 37 weeks gestation
* Birth weight ≥ 2.6 kg

Exclusion Criteria:

* Preoperative sepsis
* Preoperative renal dysfunction
* Preoperative intracranial hemorrhage
* Chromosomal abnormalities and/or genetic syndromes
* Prior intervention (catheter based or surgical)

Ages: 1 Day to 30 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2014-07; Primary Completion 2018-08-15 (Actual); Study Completion 2018-08-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chawki F Elzein, MD, Principal Investigator — Advocate Healthcare
Locations (1):
- Advocate Children's Hospital, Oak Lawn, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — http://www.advocatechildrenshospital.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Nitric Oxide on CPB: neonates receiving inhaled NO into the cardiopulmonary bypass circuit during cardiac surgery
  Inhaled Nitric Oxide: delivered inhaled Nitric Oxide into the cardiopulmonary bypass circuit during neonatal cardiac surgery
  12 patients were enrolled prospectively over 4 years period
- Control: neonates not receiving inhaled NO into the cardiopulmonary bypass
  placebo: inhaled Nitric Oxide not delivered to the cardiopulmonary bypass circuit during neonatal cardiac surgery
  12 patients were enrolled prospectively over 4 years period
Period: Overall Study
Arm/Group | Nitric Oxide on CPB | Control
Started | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nitric Oxide on CPB | Control | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 12 | 12 | 24
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: days] | 5.67 (1.87) | 5.92 (1.78) | 5.79 (1.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 9
  Male | 8 | 7 | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 3 | 5
  White | 10 | 9 | 19
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 12 | 12 | 24
anatomical diagnosis, hypoplastic left heart syndrome [Count of Participants; unit: Participants] | 10 | 11 | 21

OUTCOME MEASURES:

1. Primary Outcome: Change in Biochemical Markers of Ischemia/Reperfusion Injury and Oxidative Damage (Positive ~ Increase From Pre-op)
Description: The primary study endpoints are to evaluate whether NO delivered through the neonatal cardiopulmonary bypass (CPB) circuit can decrease various biochemical markers of ischemia/reperfusion injury and oxidative damage. Markers to be analyzed will include cardiac troponin I, interleukins (IL), tumor necrosis factor, N-terminal prohormone for brain natriuretic peptide (NT-proBNP),lactate dehydrogenase (LDH), plasma anti-oxidant levels, plasma malondialdehyde (MDA) levels.
Time Frame: Pre-op baseline and up to 12 hours after surgery
Population: Intent to treat (ITT)
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Nitric Oxide on CPB | Control
Number analyzed (Participants) | 12 | 12
ng/ml
  cardiac troponin I change | 0.46 (0.55) | 0.64 (0.64)
  IL-6 change | 11.52 (12.98) | 26.98 (27.67)
  IL-8 change | 49.36 (42.86) | 68.46 (81.09)
  TNF alpha change | 0.03 (0.20) | -0.12 (0.21)
  NT pro-BNP change | 7.03 (22.84) | 1.51 (2.29)
  LDH change | 48.85 (117.39) | 53.44 (73.58)
  Superoxide Dismutase change | -0.04 (0.04) | -0.05 (0.06)
  Plasma MDA change | 7.61 (12.90) | 10.65 (14.99)
Statistical Analysis 1: Comparison: Nitric Oxide on CPB vs Control; Null: mean cardiac troponin I changes in the NO group = mean cardiac troponin I changes in the control; Test type: Other; p > 0.05, t-test, 2 sided — This test applies to the first marker, cardiac troponin I

2. Secondary Outcome: Total Fluid Balance at 48 Hours
Description: The secondary study endpoints are to evaluate whether NO delivered through the neonatal CPB circuit can decrease the clinical signs of ischemia/reperfusion injury and/or cardiac dysfunction. Clinical parameters (post surgery) include inotropic support, fluid balances, diuretic support, ventilator times, and length of ICU stay will be evaluated.
Time Frame: 48 hours post surgery
Population: Intent to treat
Measure: Median (Inter-Quartile Range); unit: ml/kg
Arm/Group | Nitric Oxide on CPB | Control
Number analyzed (Participants) | 12 | 12
ml/kg | 32.24 [-52.90 to 165.26] | 15.93 [-160.55 to 73.245]
Statistical Analysis 1: Comparison: Nitric Oxide on CPB vs Control; Null: NO group fluid balances are the same as the control; Test type: Other; p > 0.05, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Time Until Start of Diuretic Therapy
Description: hours until start of diuretic therapy
Time Frame: Pre-op to 72 hours post surgery
Population: Intent to treat
Measure: Median (Inter-Quartile Range); unit: hour
Arm/Group | Nitric Oxide on CPB | Control
Number analyzed (Participants) | 12 | 12
hour | 25 [22.5 to 30.25] | 21.5 [19.25 to 24]

4. Secondary Outcome: Inotropic Score Day 1
Description: The Inotropic Score is an objective clinical tool used to quantify the need for cardiovascular support in children and adolescents after surgery and to predict prognosis of pediatric septic shock (higher score predicts higher risk or worse prognosis).The Inotropic Score is low if <= 20, intermediate if 21-30, and high if > 30.
  Formula used in the study:
  Daily inotropic score (mcg/kg/min) = Dopamine drip dose+ dobutamine drip dose+ (milrinone drip dose times 10) + (epinephrine drip dose times 100 )
Time Frame: 24 hours post surgery
Population: ITT
Measure: Median (Inter-Quartile Range); unit: mcg/kg/min
Arm/Group | Nitric Oxide on CPB | Control
Number analyzed (Participants) | 12 | 12
mcg/kg/min | 16.5 [12.75 to 19.75] | 15 [13.5 to 18.75]

5. Secondary Outcome: Length of Intubation and PSHU Stay
Description: Days to extubation and Pediatric Surgical Heart Unit (PSHU) length of stay (LOS) as measuring patient surgical outcomes.
Time Frame: Surgery to discharge
Population: ITT
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Nitric Oxide on CPB | Control
Number analyzed (Participants) | 12 | 12
days
  Days to extubation | 7.5 [6.25 to 9.5] | 6.5 [5.25 to 14.75]
  PSHU Length of Stay (LOS) | 15 [10.5 to 22.25] | 12 [11 to 15]

6. Other Pre Specified Outcome: Surgical Morbidity
Description: include all complications that may happen after cardiac surgery for the whole period of hospital stay, that is expected to be around 1 month. This include renal failure, prolonged intubation and ventilatory support, infections..
Time Frame: 1 month after cardiac surgery
Population: Intent to treat
Measure: Count of Participants; unit: Participants
Arm/Group | Nitric Oxide on CPB | Control
Number analyzed (Participants) | 12 | 12
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected for the entire hospitalization period, from surgical date to 104 days.
Groups:
- Nitric Oxide on CPB: Group that received nitric oxide in CPB
- Control: Group that did not receive nitric oxide in CPB
Arm/Group | Nitric Oxide on CPB | Control
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 2/12 | 1/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nitric Oxide on CPB (N=12) | Control (N=12)
Chylothorax (Blood and lymphatic system disorders) | 1 (1) | 0 (0) — chylothorax
needed cath intervention (Cardiac disorders) | 1 (1) | 1 (1) — developed narrowing at the proximal anastomosis of the Sano shunt, necessitating cardiac cath and stent implantation at the proximal Sano shunt

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-06-03): https://cdn.clinicaltrials.gov/large-docs/77/NCT02151877/Prot_SAP_000.pdf